CLINICAL TRIAL: NCT07183657
Title: Adherence to Inhaled Therapy - a Globally Overlooked Problem in Patients With Chronic Obstructive Pulmonary Disease and Bronchial Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); University Hospital Hradec Kralove (Other); University of Hradec Hralove (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NW25-09-00434
Record Dates: First submitted 2025-07-23; First posted 2025-09-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Bronchial Asthma
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Intervention; Mobile Application; Bronchial asthma; Adherence; Inhaled therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All project participants (Other): Education of inhalation technique
  Interventions: Other: Education in inhalation technique

INTERVENTIONS:
Other: Education in inhalation technique — Education in inhalation technique

SUMMARY:
Comprehensive assessment and interventions to promote adherence to inhaled therapy in patients with bronchial asthma and chronic obstructive pulmonary disease involving health care professionals caring for these patients in different settings and using the Five Steps Assessment tool and artificial intelligence methods and tools.

DETAILED DESCRIPTION:
Nonadherence to inhaled therapy is a significant problem in patients with bronchial asthma (BA) and chronic obstructive pulmonary disease (COPD), which has a negative impact on the patients´ health as well as increases the healthcare system costs. The present project focuses on multimodal assessment of adherence to inhaled therapy in patients with BA and COPD and knowledge and skills related to inhalation technique in healthcare professionals caring for patients with BA and COPD at different levels of care using our simple and validated Five Steps Assessment (FSA) tool. This is a multicenter prospective observation-interventional study planning to include 800 outpatients treated in health care facilities and nursing home residents and 200 health care professionals. During the project, a mobile/web-based app using artificial intelligence applicable to patients and healthcare professionals will be developed, implemented, and validated. Interventions (e.g., training on correct inhalation technique, educational materials, telephone/online contact, mobile/web app) to promote adherence to inhaled therapy in BA and COPD will be developed and implemented in patients. In the case of healthcare professionals, interventions (e.g., course including e-learning, mobile/web app) will be directed at increasing knowledge and skills related to inhalation technique. The impact of the interventions on patients and healthcare professionals will be verified by repeated follow-up. To be able to assess the improvement in adherence to inhaled therapy in depth, clinical and laboratory biomarkers potentially indicating the stability of COPD and BA will be measured. The outputs of the project may help to identify patients with given diagnoses at high risk of medication nonadherence and to offer simple, effective, and widely available interventions to promote medication adherence as well as to educate healthcare professionals and thereby to improve patient care.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

1. signed informed consent,
2. age ≥ 18 years,
3. previously diagnosed BA/COPD meeting GOLD 2024 and GINA 2024 diagnostic criteria,
4. ability to cooperate,
5. at least 8 weeks without exacerbation,
6. use of a particular inhaler for at least 3 months.

Exclusion Criteria:

1. pre-terminal/terminal stage of any disease,
2. uncooperative patient,
3. significant limitation of mobility or cognitive functions.

HEALTHCARE PROFESSIONALS

Inclusion Criteria:

1. signed informed consent,
2. completed education in medicine, pharmacy, or nursing,
3. more than one year of working experience,
4. care for patients taking inhaled therapy for BA/COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to inhaled treatment measured by Five Steps Assessment (FSA). | Assessment of adherence to inhaled treatment within 12 months.
  Assessment of adherence to inhaled treatment measured by patients' behavior towards inhaled treatment and a number of mistakes in inhalation technique.
Adherence to inhaled treatment measured by the Medication Adherence Report Scale (MARS). | Assessment of adherence to inhaled treatment within 12 months.
  Assessment of adherence to inhaled treatment measured by patients' behavior towards inhaled treatment and a number of mistakes in inhalation technique.
Critical knowledge measured by our own questionnaire in healthcare professionals caring for patients with COPD and bronchial asthma. | Critical knowledge related to inhalation techniques in healthcare professionals caring for patients with COPD and bronchial asthma within 12 months
  Assessment of Critical knowledge by questions on correct usage of particular inhalation systems related to inhalation techniques in healthcare professionals caring for patients with COPD and bronchial asthma.
Critical skills related to inhalation techniques measured by FSA in healthcare professionals caring for patients with COPD and bronchial asthma. | Critical skills related to inhalation techniques in healthcare professionals caring for patients with COPD and bronchial asthma within 12 months.
  Assessment of critical skills measured by a number of mistakes in inhalation technique in particular inhalation systems related to inhalation techniques in healthcare professionals caring for patients with COPD and bronchial asthma.

SECONDARY OUTCOMES:
Assessment of clinical (e.g. CAT in patients with COPD) and laboratory (e.g. white blood cell count) biomarkers potentially indicating the stability of COPD and bronchial asthma in a subgroup of patients. | Assessment of clinical and laboratory biomarkers potentially indicating the stability of COPD and bronchial asthma within 12 months.
  Changes in relevant clinical (COPD Assessment Test - CAT in patients with COPD; Asthma Control Test - ACT in patients with bronchial asthma; exacerbation frequency, and rescue medication usage) and laboratory (e.g. white blood cell count, C-reactive protein, FeNO level) biomarkers potentially indicating the stability of COPD and bronchial asthma in a subgroup of patients will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Due to sensitivity of personal and medical data of participants.

REFERENCES:
- See also: Related Info — https://portal.faf.cuni.cz/Groups/Clinical-And-Social-Pharmacy/